CLINICAL TRIAL: NCT03308071
Title: A Randomized Study Using Hypnosis for Symptom Management in Elective Orthopedic Surgery
Brief Title: Hypnosis for Symptom Management in Elective Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jessie Kittle, Clinical Instructor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-41122
Record Dates: First submitted 2017-06-23; First posted 2017-10-12 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hypnosis; Perioperative Care; Knee Arthroplasty, Total; Postoperative Pain; Postoperative Complications
Keywords: Hypnosis; Hypnotherapy; Perioperative Pain Management; Narcotic reduction; Perioperative Outcomes; Total knee replacement; Total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The treating team including surgeons, anesthesiologists, pain consultants, hospitalists who are in charge of administering pain medication and documenting outcomes will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Group (Experimental): Participants will undergo a brief hypnotic assessment, a single hypnosis session with an MD trained in hypnosis, and be given a phone number to listen to a guided self-hypnosis recording for 1 week pre-op until 2 weeks post-op.
  Interventions: Behavioral: Hypnosis
- Usual care (No Intervention): These patients will be enrolled in the study and usual care will be provided.

INTERVENTIONS:
Behavioral: Hypnosis — Hypnotic induction, relaxation, and guided imagery specific to perioperative symptoms will be administered.
  Arms: Hypnosis Group

SUMMARY:
The purpose of the study is to determine if teaching self-hypnosis techniques to patients prior to knee replacement surgery will decrease their pain medication requirements, pain medication side-effects, length of stay in the hospital, readmission rates, pain, anxiety, physical function, satisfaction scores, and cost of admission.

DETAILED DESCRIPTION:
Patients will be recruited by through orthopedic surgery clinics or contacted by after pre-screening via chart review and given an information brochure. If they are interested in the trial will be emailed or given a paper copy of the consent form and scheduled for a single additional visit in the Integrative Medicine Center at Hoover Pavilion approximately 1 week before surgery. At the single study visit, participants would be consented, then a mini-mental state test would be performed to determine if participants are eligible by a score of 25 or above. If eligible, participants would be asked to fill out surveys relating to demographics, attitudes and experience with hypnosis, and detailed pain medication usage. Then, participants would be randomized to hypnosis vs. no hypnosis. The hypnosis group will undergo a Hypnotic Induction Profile to score hypnotizability, then be lead through a hypnosis induction and read a perioperative symptom management script, then re-alerted from hypnosis. Patients in this group would then be asked to listen to the same hypnosis script on a telephone recording twice per day until after the surgery when participants feel they don't need it anymore.

The control group will fill out the surveys and the study visit will end. Participants will be asked not to use any hypnosis until the trial period is over. Data regarding pain, activity, and satisfaction is already collected by email survey or by Ipad in orthopedic clinic at or before the pre-op visit, and 3 months post-op.

Patients in the knee study will be asked to fill out the same surveys around the two week and six week post-op orthopedic clinic visits as well. One additional survey will be added at the 2 week post-op visit to reassess attitudes and experience with hypnosis, and detailed pain medication usage. Those participants who do not fill out the survey will be called and/or emailed to remind them to fill it out.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* scheduled for a primary, unilateral, total knee replacement surgery within the study period
* able to commit to a single study clinic visit at least one week prior to their scheduled surgery and use of phone recordings
* able to read and understand English
* Score at least 25 on mini-mental state exam

Exclusion Criteria:

* severe psychiatric or structural brain disease (ie. psychosis, stroke with functional impairment, dementia)
* current use of hypnosis/self-hypnosis
* enrolled in other clinical trials related to pain management or length of stay
* hearing impairment that would impede ability to listen to a phone recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Narcotic use | Index hospitalization for total knee replacement, average 2-3 days
  Total narcotic use during the hospital stay will be calculated in "morphine equivalents"

SECONDARY OUTCOMES:
Narcotic prescriptions | 1 month before, and 3 months and 1 year after joint replacement
  Total narcotics prescribed in the outpatient setting
Narcotic-associated side effects | Index hospitalization for total knee replacement, average 2-3 days
  Incidence of delirium, constipation, urinary retention, respiratory depression
UCLA activity scores | At the pre-op visit with the surgeon and 2, 6 and 12 weeks post-op
  Classifies the activity level of joint replacement patients
KOOS Jr Survey | At the pre-op visit with the surgeon and 2, 6 and 12 weeks post-op
  Knee injury and osteoarthritis outcome score
VR-12 Survey | At the pre-op visit with the surgeon and 2, 6 and 12 weeks post-op
  Measures health-related quality of life
Knee Society Score | At the pre-op visit with the surgeon and 12 weeks post-op
  Prosthesis function and patients' functional abilities after total knee arthroplasty (TKA)
Number of days hospitalized | Reported once , after patient is discharged (1 day)
  Total number of days hospitalized for total knee replacement surgery
Satisfaction with hypnosis survey | Pre-op and 2 weeks post-op
  Attitudes and expectations regarding hypnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University/Stanford Healthcare, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Markovits J, Blaha O, Zhao E, Spiegel D. Effects of hypnosis versus enhanced standard of care on postoperative opioid use after total knee arthroplasty: the HYPNO-TKA randomized clinical trial. Reg Anesth Pain Med. 2022 Jun 17:rapm-2022-103493. doi: 10.1136/rapm-2022-103493. Online ahead of print. PMID 35715013